CLINICAL TRIAL: NCT02379637
Title: A Randomized, Parallel-Group, Double-Blind, Placebo-Controlled, Multiple-Dose, Proof-of-Concept Study to Evaluate the Efficacy of N-acetylcysteine Capsules in the Treatment of the Common Cold (Viral URTI) Associated With Cough in an Adult Population
Brief Title: Study to Evaluate the Efficacy of N-acetylcysteine (NAC) in the Treatment of the Common Cold and Cough
Acronym: NAC cold cough
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2160-A-201
Record Dates: First submitted 2015-02-13; First posted 2015-03-05 (Estimated); Results first posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-05

CONDITIONS: Common Cold Associated With Cough
Keywords: N-acetylcysteine; adults; cough and cold
MeSH Terms: conditions — Cough; Common Cold | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A N-acetylcysteine (Experimental): N-acetylcysteine
  Interventions: Drug: N-acetylcysteine
- B Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-acetylcysteine
  Arms: A N-acetylcysteine
Drug: Placebo
  Arms: B Placebo

SUMMARY:
This study is designed to improve knowledge regarding the initial effectiveness of N-acetylcysteine (NAC) on cold and cough symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Cold/URTI symptoms occurring no more than 4 days
* cough due to a cold or acute viral (URTI) with an onset of no more than 3 days
* cough frequency with specified cut-off

Exclusion Criteria:

* A subchronic, or chronic cough (cough duration > 2 months) due to any condition other than a cold/URTI
* Diagnosed as suffering from any pulmonary conditions associated with cough, e.g., chronic obstructive pulmonary disease (COPD), acute or chronic bronchitis, asthma, cystic fibrosis
* Taking any medications known to induce cough
* Fever of greater than 39°C (102°F) orally
* Complication of the common cold like otitis media, severe sinusitis, or pneumonia
* Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- Canada (5):
  - Chicoutimi, Quebec
  - Montreal, Quebec
  - Québec, Quebec
  - Sherbrook, Quebec
  - Victoriaville, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 8 centers in canada Start date 26 Jan 2015 End date 01 Apr 2015
Pre-assignment Details: Screening and randomization are on day 1 Duration of the study = 7 days
Groups:
- A N-acetylcysteine: N-acetylcysteine
  N-acetylcysteine, capsules, 800 mg 3 times daily
- B Placebo: Placebo
  Placebo, matching capsules three times daily
Period: Overall Study
Arm/Group | A N-acetylcysteine | B Placebo
Started | 35 | 35
Completed | 33 | 34
Not Completed | 2 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A N-acetylcysteine | B Placebo | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (11.06) | 34 (12.9) | 33.5 (11.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 46
  Male | 12 | 12 | 24
Region of Enrollment [Number; unit: participants]
  Canada | 35 | 35 | 70
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 26.3 (4.49) | 27.3 (4.59) | 26.8 (4.53)

OUTCOME MEASURES:

1. Primary Outcome: Cough Count (Number of Coughs Will be Measured by a 24-hour Ambulatory Cough Monitoring System for the First 72 Hours)
Description: Number of coughs will be measured by a 24-hour ambulatory cough monitoring system for the first 72 hours
Time Frame: 72 hours
Population: Full Analysis set
Measure: Mean (Standard Deviation); unit: log-transformed total cough count
Arm/Group | A N-acetylcysteine | B Placebo
Number analyzed (Participants) | 35 | 35
log-transformed total cough count | 6.92 (0.95) | 6.51 (0.83)

2. Secondary Outcome: Safety of Daily Dose of NAC (Number of Patients With Adverse Advents)
Description: Number of patients with adverse advents
Time Frame: 7 Days
Measure: Number; unit: participants
Arm/Group | A N-acetylcysteine | B Placebo
Number analyzed (Participants) | 35 | 35
participants | 4 | 4

ADVERSE EVENTS:
Arm/Group | A N-acetylcysteine | B Placebo
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 2/35 | 2/35
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A N-acetylcysteine (N=35) | B Placebo (N=35)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor shall review results communications prior to public release to evaluate the manuscript for accuracy, ascertain whether information (other than the results of the Clinical Trial) is being improperly disclosed, provided information which may have not have yet been made available by the Sponsor, provide input for consideration regarding the content and/or conclusion(s) of the manuscript and determine whether the manuscript discloses any potentially patentable invention(s).